CLINICAL TRIAL: NCT05589688
Title: Individualization of Dosage Regimens in Obese Patients: Application to Acyclovir
Acronym: ACICLOPTIM
Status: Recruiting | Phase: Phase 1 | Type: Interventional
Sponsor: University Hospital, Toulouse (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: RC31/21/0610
Record Dates: First submitted 2022-10-17; First posted 2022-10-21 (Actual); Last update posted 2025-12-31 (Actual); Status verified 2025-12

CONDITIONS: Obesity
MeSH Terms: conditions — Obesity | interventions — Acyclovir

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- acyclovir (Experimental): Subjects take a single dose of 5 mg/kg infused over 1 hour.
  Interventions: Drug: Acyclovir

INTERVENTIONS:
Drug: Acyclovir — Subjects will receive a single dose of 5 mg/kg infused over 1 hour. Then, 13 blood samples after placement of a catheter, and 4 urine samples will be taken over the 12 hours following the start of administration

SUMMARY:
The number of obese people will reach 50% of the world population by 2035. Obesity is a chronic disease. For obese patients, dosage regimens have been determined for patients with a "normal" BMI between 20-30 kg/m2. Based on plasma and urine concentrations, a pharmacokinetic model will be performed to study in healthy volunteers, the predictive character of lean mass, measured by DEXA, on renal elimination and therefore on acyclovir exposure. The main objective of this study is to evaluate, in 4 volunteers groups representative of (1) non-obese (18-24.9 kg/m2), (2) overweight (25-29.9 kg/m2), (3) grade 1 obesity (30-34.9 kg/m2) and (4) grade 2 obesity (35-39.9 kg/m2), the predictive nature of lean mass, measured by DEXA, on renal elimination and therefore on acyclovir exposure.

DETAILED DESCRIPTION:
This study will complement the clinical data on acyclovir in healthy volunteers considering that current knowledge in terms of drugs use in obese subjects is not sufficient to guarantee the efficacy and/or toxicity absence of exposure. As a consequence, this lack of certainties leads physicians to propose dosages without exceeding a threshold defined according to (i) their experience, (ii) data obtained for BMI < 30 kg/m2 and/or (iii) an approximate criterion derived from the total weight (adjusted weight...). Acyclovir is a systemic antiviral drug indicated for the treatment of Herpes Simplex virus (HSV) and Varicella Zoster (VZV) mucosal infections at 15 mg/kg/d in three divided doses, or more severe infections (e.g., herpetic meningoencephalitis) at higher dosage regimen (30 to 45 mg/kg/d in three divided doses).

ELIGIBILITY:
Inclusion Criteria:

* healthy volunteers with a BMI between 18 and 39,9 kg/m2, divided into 4 groups: 5 non-obese volunteers (BMI between 18 and 24,9 kg/m2), 5 overweight volunteers (BMI between 25 and 29,9 kg/m2), 5 volunteers with grade 1 obesity (BMI between 30 and 34,9 kg/m2) and 5 volunteers with grade 2 obesity (BMI between 35 and 39,9 kg/m2),
* volunteers with a aGFR > 50 ml/min,
* with a good venous pathway for kinetics,
* women on contraception or postmenopausal women,
* person who has given written consent and affiliated with the public health insurance.

Exclusion Criteria:

* volunteers with nephrotoxic co-prescriptions and/or co-prescriptions that would modify the pharmacokinetics of acyclovir like diuretics, NSAIDs or statins,
* having presented serious allergies to a drug (e.g. angioedema...), with large parenchyma insufficiencies (e.g., hepatic insufficiency, heart failure...),
* with diabetes or taking anti-diabetics due to the possible deterioration of renal function in diabetic patients,
* with arterial hypertension or taking antihypertensive drugs due to the possible modification of renal clearance by modification of blood flow,
* drug interactions with acyclovir (H2 receptor antagonists (e.g., Cimetidine), Probenecid, Mycophenolate Mofetil, Lithium, Anti-calcineurins (Ciclosporin, Tacrolimus)),
* volunteers taking anticoagulants,
* hypersensitivity to acyclovir,
* pregnant woman,
* participation in another clinical study in the last two months
* volunteers with ongoing viral HSV/VZV infection treated with acyclovir,
* adults under guardianship or other legal protection, deprived of their liberty by judicial or administrative decision

Ages: 18 Years to 50 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 20 (Estimated)
Dates: Start 2024-04-09 (Actual); Primary Completion 2026-12 (Estimated); Study Completion 2026-12 (Estimated)

PRIMARY OUTCOMES:
Renal elimination clearance | Day 1
  To quantify the relationship between lean body mass, measured by Dual-energy x-ray absorptiometry (DEXA), and the true absolute glomerular filtration rate (GFRa) which is estimated by the renal elimination clearance of acyclovir.

SECONDARY OUTCOMES:
the interindividual variability of acyclovir exposure : lean mass | Day 1
  To measure lean mass by DEXA on subjects
the interindividual variability of acyclovir exposure : glomerular filtration rate | Day 1
  A blood sample will be taken for this purpose to assess the renal function of the volunteer by measuring his uremia and his creatinine allowing the calculation of the glomerular filtration rate.
the qualitative compilation of adverse events associated with acyclovir infusion observed and reported by the volunteer. | Day 1, Day 2
  adverse events reported by volunteers

CONTACTS AND LOCATIONS:
Overall Officials: Sarah Baklouti, PharmD, Principal Investigator — University Hospital, Toulouse
Locations (1):
- Toulouse Hospital, Toulouse, France

IPD SHARING:
Plan to Share IPD: No